CLINICAL TRIAL: NCT07126093
Title: An Exploratory Study on the Application of Focal High-intensity Focused Ultrasound (HIFU) Therapy Combined With Systemic Novel Hormone Therapy in Advanced Prostate Cancer
Brief Title: High-intensity Focused Ultrasound Combined With Novel Hormone Therapy in Advanced Prostate Cancer
Acronym: HIFU NHT PCa
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Zhang Yu, Attending Physician and assistant resarcher, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HIFUNHT20250808
Record Dates: First submitted 2025-08-08; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; HIFU; NHT
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined group (Experimental): Participants in this arm will receive HIFU combined with standard NHT therapy
  Interventions: Combination Product: focal high-intensity focused ultrasound therapy combined with standard novel hormonal therapy
- Standard treatment group (Other): Participants in this arm will receive standard NHT
  Interventions: Other: Standard novel hormonal therapy only

INTERVENTIONS:
Combination Product: focal high-intensity focused ultrasound therapy combined with standard novel hormonal therapy — The participants in the intervention arm will receive HIFU combined with standard NHT. Depending on the location of the lesion, tumor load and the pathological conditions, hemicglandular ablation or focal ablation was selectively administered. The safe boundary was set at 3mm, with a power of 300W and a pulse width of 30ms. Novel endocrine therapy was given after HIFU treatment
  Arms: Combined group
Other: Standard novel hormonal therapy only — Participants in the control arm will receive standard NHT.
  Arms: Standard treatment group

SUMMARY:
The goal of this clinical trial is to explore the feasibility and the synergistic anti-cancer effect of high-intensity focused ultrasound (HIFU) combined with novel hormone therapy (NHT) in advanced prostate cancer (PCa). The main questions it aims to answer are: (1) whether could HIFU combined with NHT improve the long-term survival of patients with advanced PCa and alleviate local symptoms? (2) Does the synergistic effect of HIFU combined with NHT exist? Researchers will compare HIFU combined with NHT to NHT alone in advanced PCa patients. Participants will receive HIFU before NHT therapy or only receive NHT. In addition, participants are encouraged to record local symptoms condition and conduct regular follow-up.

DETAILED DESCRIPTION:
An RCT study is conducted to include patients with advanced prostate cancer, who are randomly divided into two groups: the NHT alone group and the HIFU combined with NHT group. We compare the PFS after treatment to explore whether HIFU plus NHT improve the long-term survival and postpone progression. All patients will sign the informed consent form before enrollment and will be taken good care during study period. Patients will be screened according to the inclusion and exclusion criteria and will be given therapy according to randomization. Research data will be analyzed by a professional statistics team. The completion of the research will facilitate the expansion of HIFU into the comprehensive treatment of advanced PCa and will help improve the survival of such patients.

ELIGIBILITY:
Inclusion Criteria:

1. Male patients who are at least 18 years old;
2. The physical condition score of the Eastern Cooperative Oncology Group (ECOG) in the United States is 0 to 2 points.
3. Newly diagnosed patients with advanced prostate cancer confirmed by PSMA PET/CT (including metastatic hormone-sensitive prostate cancer or inoperable locally advanced prostate cancer);
4. No previous treatments for prostate cancer have been received;
5. After assessment, there was no obvious insufficiency of vital organs.
6. Sign the written informed consent form for this study, indicating that they fully understand the purpose and process of this study and are willing to participate in it.

Exclusion Criteria:

1. A history of any other active malignant tumor within 2 years (excluding well-treated basal cell or squamous cell skin cancer, superficial bladder cancer, or any other carcinoma in situ currently in complete remission);
2. Prostate biopsy pathology shows sarcomatoid cells, intraductal carcinoma, and neuroendocrine cell components;
3. Accompanied by severe comorbidities, immunosuppression, severe mental illness, severe activity limitation and other conditions that prevent compliance with clinical trials;
4. Currently participating in other clinical trials related to this disease;
5. According to the researcher's judgment, there are relevant evaluations that do not align with the best interests of the subjects' participation in the study (such as affecting the subjects' sense of happiness) or may hinder, restrict or interfere with the research protocol;
6. Concurrent infectious diseases that affect the treatment outcome.

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2029-10-31 (Estimated); Study Completion 2030-10-31 (Estimated)

PRIMARY OUTCOMES:
progression-free survival (PFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 80 months
  PFS refers to the time from the start of randomization to disease progression. Disease progression includes biochemical progression, clinical progression and imaging progression. Biochemical progression is defined as a PSA increase of more than 25% and an absolute increase of 2ng/ml compared to the baseline/minimum value. The definition of clinical progression is the emergence of any new clinical symptoms related to the primary disease and metastases of prostate cancer. The definition of imaging progression in imaging is the appearance of any new metastatic lesions.

SECONDARY OUTCOMES:
overall survival (OS) | From date of randomization until the date of death from any cause, assessed up to 80 months
  It refers to the time from the start of randomization to death for any reason
Time to castration resistance | the time from the start of randomization to the occurrence of castration resistance, assessed up to 80 months
  Castration resistance is defined as : serum testosterone <50 ng/dL or 1.7 nmol/L plus any one of the following: ① Biochemical progression: Three consecutive increases in PSA (at least one week apart), with two increases of 50% compared to the lowest value, and the absolute value >2 ng/mL; ② Radiological progress: Two or more new bone metastases are found in imaging examinations such as bone scans, PET/CT, or one or more soft tissue lesions evaluated by the solid tumor response assessment criteria (RECIST 1.1 criteria, Appendix 1);

IPD SHARING:
Plan to Share IPD: No
While supporting data sharing principles, individual participant data (IPD) from this trial cannot be shared due to its proprietary nature and the need to protect individual information and intellectual property. Aggregate results will be published according to regulatory requirements and made available through standard reporting channels.